CLINICAL TRIAL: NCT00664430
Title: Efficacy and Safety of Paricalcitol on the Treatment of Secondary Hyperparathyroidism in Calcitriol Resistant Dialysis Subjects
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment rate
Sponsor: Abbott (Industry)
Collaborators: Statistika Consultoria Ltda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W10-131
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Results first posted 2010-08-18 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Secondary Hyperparathyroidism; Dialysis
Keywords: Dialysis; Calcitriol Resistant; Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — Calcitriol; paricalcitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Calcitriol challenge followed by paricalcitol (Other): Participants began a controlled calcitriol therapy period (calcitriol challenge) to confirm calcitriol resistance. After this period, those who failed to reduce PTH (according to parameters in protocol) initiated paricalcitol therapy.
  Interventions: Drug: Calcitriol; Drug: Paricalcitol

INTERVENTIONS:
Drug: Calcitriol — Initial doses determined according to the National Kidney Foundation's Kidney Disease Outcomes Quality Initiative (KDOQI) guideline (Am J Kidney Dis 2003;42(4)Suppl 3:S1-S201). During therapy, calcitriol dose may be modified by 0.5 - 1 mcg at 2- to 4-week intervals.
  Other Names: Calcijex
Drug: Paricalcitol — Dose calculated by 0.04 to 0.1 microgram per kilogram (mcg/kg). Paricalcitol will be administered intravenously after the participants' dialysis. The paricalcitol dose will be titrated every 2 weeks until iPTH presents a reduction or up to 4 months, after which it will be adjusted monthly based on serum PTH, calcium, phosphorus and albumin measurements. Dosing may be modified by 2-4 mcg increments at 2- to 4-week intervals.
  Other Names: ABT-358; Zemplar; Paracalcitol

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of paricalcitol in participants with moderate to severe secondary hyperparathyroidism (SHPT) undergoing hemodialysis who are resistant to treatment with calcitriol.

DETAILED DESCRIPTION:
This is a multi-center, prospective, open label, one arm, phase IV study designed to demonstrate paricalcitol efficacy and safety in the treatment of moderate to severe secondary hyperparathyroidism in calcitriol resistant participants on dialysis.

Following screening, participants began an 8-week controlled calcitriol therapy period. Participants whose parathyroid hormone (PTH) levels decreased were to be discontinued from the study. Those whose PTH levels did not decrease began paricalcitol therapy using a dose calculated by 0.04 to 0.1 microgram per kilogram (mcg/kg). Paricalcitol was administered intravenously at anytime during the subjects' dialysis. The paricalcitol dose was to be titrated every 2 weeks until iPTH was reduced or up to 4 months, after which it was to be adjusted monthly for 1 year based on serum PTH, calcium, phosphorus, and albumin measurements.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants > 18 years of age, with chronic kidney disease (CKD) stage V;
* Participants with diagnosis of calcitriol resistance defined as: Episodes of hypercalcemia and/or hyperphosphatemia (defined as an episode of calcium or phosphorus above Upper Limit of Normal or documented by medical history stating that the treatment with calcitriol was discontinued due to hypercalcemia and/or hyperphosphatemia) that precludes treatment continuation and/or persistent PTH above 600pg/mL during the calcitriol therapy;
* PTH value at screening visit between 600 pg/mL and 2,000 pg/mL;
* Stable clinical conditions;
* Participant has voluntarily consented to participate in the study, by signing and dating an informed consent form, approved by an Institutional Review Board (IRB)/Independent Ethics Committee (IEC), after the nature of the study has been explained and all his questions about the study have been elucidated. The informed consent must be signed before any study-specific procedures are performed.

Exclusion Criteria:

* Previous parathyroidectomy;
* Presence of hypercalcemia (corrected Ca > 10.5 mg/dL) and/or hyperphosphatemia (P > 6.0 mg/dL) and/or Ca x P product > 60, at screening visit (corrected Ca calculated by: [4 - participant's serum albumin (g/dL)] x 0.8 + participant's serum Ca value);
* Severe and/or unstable clinical conditions, e.g., congestive heart failure, advanced cancer, advanced HIV disease, severe endocrinopathies, uncompensated diabetes mellitus, life-threatening cardiac arrhythmias, etc;
* Abnormal liver tests (> 1.5 times above upper limit of normal);
* Pregnant or breast-feeding women;
* Evidence of vitamin D toxicity;
* Known hypersensitivity to any study drug components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-01; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lino Rodrigues, MD, Study Director — Abbott
Locations (2):
- Brazil (2):
  - Site Reference ID/Investigator# 7118, São Paulo
  - Site Reference ID/Investigator# 7114, São Paulo

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After Screening, participants entered an 8-week controlled calcitriol period. Participants whose parathyroid hormone (PTH) levels decreased after 8 weeks (i.e., participants who were not resistant to calcitriol) were discontinued from the study.
Groups:
- Calcitriol Challenge Followed by Paricalcitol: To confirm this resistance, participants began a controlled calcitriol therapy period. After this period, participants whose parathyroid hormone (PTH) levels were not reduced according to parameters in protocol were to begin a paricalcitol titration period of up to 4 months, followed by paricalcitol therapy for up to 1 year.
Period: Overall Study
Arm/Group | Calcitriol Challenge Followed by Paricalcitol
Started | 13
Completed | 0 (Study terminated early due to low enrollment rate.)
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | Calcitriol Challenge Followed by Paricalcitol
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Region of Enrollment [Number; unit: participants]
  Brazil | 13

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With a 50% Reduction in Parathyroid Hormone (PTH) Levels Relative to Visit 4 Values
Description: This outcome was measured at Visit 15, which could occur at different timepoints from study start, depending on the duration of each study period for each participant, relative to values on Visit 4. For participants who did not perform visit 4, the reduction of the PTH levels were to be assessed relative to visit 5 values.
Time Frame: Up to Week 24
Population: No efficacy analysis was performed in this study. At the time the study was stopped, 3 participants were receiving paricalcitol, but none of them had reached the time point for the primary analysis.
Measure: Number; unit: Proportion of participants
Arm/Group | Calcitriol Challenge Followed by Paricalcitol
Number analyzed (Participants) | 0

2. Secondary Outcome: Changes in Bone Remodeling Markers Over Time
Description: Deoxypyridinoline and bone-specific alkaline phosphatase levels were to be measured every 3 months and changes over time analyzed using descriptive statistics.
Time Frame: Every 3 months
Population: No efficacy analysis was performed in this study. At the time the study was stopped, 3 participants were receiving paricalcitol, but none of them had reached the time point for the secondary analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Calcitriol Challenge Followed by Paricalcitol
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Adverse Events
Description: The occurrence of adverse events was considered a secondary endpoint in this study. For details on adverse events that occurred prior to study termination, refer to the safety section below.
Time Frame: Up to 1 year
Measure: Number; unit: Participants
Arm/Group | Calcitriol Challenge Followed by Paricalcitol
Number analyzed (Participants) | 13
Participants | 3

ADVERSE EVENTS:
Arm/Group | Calcitriol Challenge Followed by Paricalcitol
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 3/13
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calcitriol Challenge Followed by Paricalcitol (N=13)
Headache (Nervous system disorders) | 2 (5)
Tachycardia (Cardiac disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (3)
Hypotension (Vascular disorders) | 1 (1)
Transitory dyspepsia (Gastrointestinal disorders) | 1 (1)
Paresthesia of right upper limbs (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to no efficacy evaluation. All adverse events occurred during calcitriol challenge phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.